CLINICAL TRIAL: NCT00120991
Title: Off-Pump Coronary Artery Bypass Grafting Versus Conventional Coronary Artery Bypass Grafting on Postoperative Mortality and Morbidity, A Randomized Clinical Trial
Brief Title: Best Bypass Surgery (BBS) Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Heart Foundation (Other); The Danish Medical Research Council (Other); Copenhagen Hospital Corporation (Other)
Responsible Party: Dept Cardiothorax Surgery, Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2001-11-DP-83-RKF-22
Record Dates: First submitted 2005-07-08; First posted 2005-07-19 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Heart Disease; Cardiovascular Disease
Keywords: Coronary artery bypass grafting; OPCAB
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases | interventions — Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Procedure: Coronary artery bypass grafting

SUMMARY:
There is evidence linking cardiopulmonary bypass to negative side effects when used for coronary artery bypass grafting. Coronary artery bypass grafting can be performed without the use of cardiopulmonary bypass. The purpose of this study is to determine the positive and negative effects of coronary artery bypass grafting with or without the use of cardiopulmonary bypass. The patients will be followed at least one year after surgery.

DETAILED DESCRIPTION:
Objectives:

To evaluate the beneficial and harmful effects of off-pump coronary artery bypass grafting (OPCAB) versus conventional coronary artery bypass grafting (CCABG) using a heart- and lung machine in patients with three-vessel coronary artery disease.

Trial population:

Consecutive patients > 54 years of age with three-vessel coronary artery disease with EuroSCORE of 5-16 undergoing elective or sub-acute coronary artery bypass grafting, giving written informed consent, and where randomisation can be accomplished preoperatively. The study will include 330 patients.

Trial design:

The Best Bypass Surgery Trial (BBS Trial) is a randomised trial. Patients will be randomised to one of two groups. The randomisation will be 1:1, in blocks, stratified by gender, age (55 to 65 years; > 65 years), diabetes mellitus, and EuroSCORE (5-7; 8-10; 11-13; 14-16). The patients will be randomised to OPCAB surgery or CCABG surgery.

The interventions:

In the OPCAB group, the revascularization procedure will be performed on the beating heart with a stabilizer to demobilize the target coronary arteries. When access is needed for posterior coronary arteries a suction device will lift the heart. In the CCABG group, the revascularization procedure will be performed with the use of a heart- and lung machine in normothermia, aortic cross clamp, and with cold cardioplegic arrest. In both groups, the left internal mammary artery and saphenous vein grafts are standard graft material.

Outcome measures:

The aim of the study is to examine the value of OPCAB revascularization compared to CCABG revascularization on the following outcome measures:

* Primary: The composite outcome measure of mortality (of all causes), acute myocardial infarction, cardiac arrest with successful resuscitation, low cardiac output syndrome, or major neurological deficit.
* Secondary: Hyper dynamic shock; atrial fibrillation, respiratory insufficiency requiring intubation >24 hours , need for pacing > 1 day due to 2º AV-blockage or nodal rhythm; renal complications, i.e., serum creatinine > 200 μmol/l, or need for acute dialysis; re-operation for bleeding, pneumonia; serious adverse events; duration of stay in intensive care unit; duration of stay in the hospital; quality of life after 3 and 12 month; graft patency at one year postoperatively defined by coronary angiography. In addition, cognitive function will be assessed after three and 12 months in the first 120 patients randomized.

ELIGIBILITY:
Inclusion Criteria:

* Known ischemic three vessel heart disease affecting one of the marginal coronary arteries
* Age > 54 years
* Scheduled for elective or subacute CABG
* EuroSCORE > 4 and < 17
* The patient has signed written informed consent before randomization and surgery.

Exclusion Criteria:

* Previous heart surgery
* Ejection fraction < 30 %
* Unstable preoperative condition, i.e., continuous infusion of inotropics on the day of the operation
* Patient unable to give informed consent.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2002-04; Primary Completion 2006-03 (Actual); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | Short and long term
Acute myocardial infarction
Cardiac arrest with successful resuscitation
Low cardiac output syndrome/cardiogenic shock
Stroke
Need for renewed cardiac revascularization procedure

SECONDARY OUTCOMES:
Hyper dynamic shock
Atrial fibrillation during index admission
Need for pacing > 24 hours
Renal complications, i.e., increased serum creatinine
Reoperation for bleeding during index admission
Pneumonia
Respiratory insufficiency requiring intubation > 24 hours postoperatively
Serious adverse events
Duration of stay in intensive care unit
Duration of stay in the hospital
Quality of life after 3 and 12 month
Graft patency at one year postoperatively defined by coronary angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Christian H. Møller, MD, Principal Investigator — Dept. of Cardiothoracic Surgery and Copenhagen Trial Unit, Rigshospitalet, Copenhagen; Daniel A. Steinbrüchel, Professor, Study Director — Dept. of Cardiothoracic Surgery, Rigshospitalet, Copenhagen; Christian Gluud, Consultant, Study Chair — Copenhagen Trial Unit, Rigshospitalet, Copenhagen; Jan K. Madsen, Consultant, Study Chair — Dept. of Cardiology, Amtssygehuset i Gentofte, Copenhagen
Locations (1):
- Dept. Cardiothoracic Surgery, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Moller CH, Perko MJ, Lund JT, Andersen LW, Kelbaek H, Madsen JK, Winkel P, Gluud C, Steinbruchel DA. Three-year follow-up in a subset of high-risk patients randomly assigned to off-pump versus on-pump coronary artery bypass surgery: the Best Bypass Surgery trial. Heart. 2011 Jun;97(11):907-13. doi: 10.1136/hrt.2010.211680. Epub 2011 Mar 17. PMID 21415073
- [Derived] Moller CH, Perko MJ, Lund JT, Andersen LW, Kelbaek H, Madsen JK, Winkel P, Gluud C, Steinbruchel DA. No major differences in 30-day outcomes in high-risk patients randomized to off-pump versus on-pump coronary bypass surgery: the best bypass surgery trial. Circulation. 2010 Feb 2;121(4):498-504. doi: 10.1161/CIRCULATIONAHA.109.880443. Epub 2010 Jan 18. PMID 20083683
- [Derived] Jensen BO, Rasmussen LS, Steinbruchel DA. Cognitive outcomes in elderly high-risk patients 1 year after off-pump versus on-pump coronary artery bypass grafting. A randomized trial. Eur J Cardiothorac Surg. 2008 Nov;34(5):1016-21. doi: 10.1016/j.ejcts.2008.07.053. Epub 2008 Sep 7. PMID 18778948